CLINICAL TRIAL: NCT03437005
Title: Alterations in the Human Microbiome With Commonly Used Topical Medications
Brief Title: Alternation in the Human Microbiome With Commonly Used Topical Medications
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 390406
Record Dates: First submitted 2018-02-12; First posted 2018-02-19 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-02

CONDITIONS: Healthy
Keywords: Human microbiome; Topical; Steroid; Anti-fungal

STUDY DESIGN:
Intervention Model Description: The patient will be randomized to one of two groups, with one group receiving ketoconazole cream and the other receiving desonide ointment.
Who Masked: Participant, Investigator
Masking Description: Investigator and subject will be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Desonide 0.05% (Experimental): Low potency steroid topical medication applied to specific locations on the face and extremities, twice daily for two weeks
  Interventions: Drug: Desonide 0.05%
- Ketoconazole 2% (Experimental): Antifungal topical medication applied to specific locations on the face and extremities, twice daily for two weeks
  Interventions: Drug: Ketoconazole 2%

INTERVENTIONS:
Drug: Desonide 0.05% — Desonide 0.05% ointment topically twice daily for two weeks
  Arms: Desonide 0.05%
Drug: Ketoconazole 2% — Ketoconazole 2% cream topically twice daily for two weeks
  Arms: Ketoconazole 2%

SUMMARY:
The global aim of this study is to investigate how the human microbiome changes from baseline with commonly used topical medications such as topical antifungals, low to mid potency topical steroids and emollients.

The specific aims are as follows:

1. Investigate whether ketoconazole cream, a commonly used topical antifungal, causes alterations in the human skin microbiome with short-term use.
2. Investigate whether desonide 0.05 % ointment, a commonly used low potency topical steroid, alters the human microbiome with short-term use.

DETAILED DESCRIPTION:
The microorganisms present on human skin influence human health and disease. Older methods of studying the skin microbiota, such as culture based techniques, favored bacteria, which readily grew under standard laboratory conditions, compared to current molecular approaches, which have shown a greater diversity of skin microbiota. Human skin is a large organ that contains a wide range of physiological and topographical diversity. Distinct niches exist which predispose certain areas, such as hairy, moist underarms to a different bacterial community from dry, smooth sites, such as forearms. Given that the skin is a critical barrier between the body's internal environment and the external environment, characterization of the microbiota of the skin may provide insight into the balance between skin health and disease.

Certain inflammatory skin diseases, such as seborrheic dermatitis, atopic dermatitis and psoriasis, have characteristic sites of involvement. The NIH funded Human Microbiome Project (HMP) aims to characterize the human microbiota and its role in health and disease. Recent research by the HMP showed that certain sites, such as the antecubital and popliteal fossa, sites commonly affected in atopic dermatitis, shared similar groups of organisms and distinct microbial communities. Sebaceous sites, commonly affected in seborrheic dermatitis, also shared similar microbial communities. In addition, Kong et al., showed that changes in microbial communities were temporally associated with disease flares in atopic dermatitis patients. Changes in the microbial communities in atopic dermatitis patients were not only associated with disease flares, but were also associated with whether the patient received treatment with topical medications, including antimicrobial or anti-inflammatory medications, during flares. These findings suggest that communities of microbes are important in the initiation and perpetuation of certain skin diseases and that the topical medications used in treatment of these diseases have an important role, which may be related to their alteration of the microbiome.

The most commonly used treatments in dermatology include topical steroids and topical antifungals, which have long established safety and efficacy. Understanding the changes that these topical medications cause in the human microbiome will provide further insight into their role in the treatment of certain skin diseases and may assist us in developing new therapies in the future.

ELIGIBILITY:
The inclusion criteria:

• Adults at least 18 years of age.

The exclusion criteria:

* Individuals with known chronically active skin diseases, including atopic dermatitis, psoriasis, seborrheic dermatitis, other autoimmune and inflammatory skin conditions.

  * Patients with a history of skin cancer, multiple nevi, or other isolated lesions will not be excluded.
* Individuals who have used topical, intravenous, intramuscular, or oral antibiotics within the last 6 months
* Individuals with known allergies to any of the study medications.
* Individuals younger than 18 years of age.
* Adults unable to consent
* Non-English speaking individuals. Given the complexity in the instructions that subjects will need to follow for proper sample collection, we will not seek to recruit non-English speaking individuals for this pilot study.
* Prisoners

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2013-01-28 (Actual); Primary Completion 2026-09-28 (Estimated); Study Completion 2026-09-28 (Estimated)

PRIMARY OUTCOMES:
Number of bacteria per each species | 2 weeks after initial dispensing
  Percentage of various bacteria present on each skin site

SECONDARY OUTCOMES:
Number of species at test sites | 2 weeks after initial dispensing
  The taxonomic diversity and evenness of each skin site's microbiome

CONTACTS AND LOCATIONS:
Overall Officials: Emanual Maverakis, MD, Principal Investigator — UC Davis
Locations (1):
- University of California, Davis, Department of Dermatology, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: No